CLINICAL TRIAL: NCT04188704
Title: Comparative Study of the Inclination Angle and Complications of Eccentric Grafts Position in ACL Reconstruction and Normal ACL: Retrospective Cohort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Collaborators: Thammasat University (Other)
Responsible Party: Principal Investigator, Jatupon Kongtharvonskul, principle investigator, Ramathibodi Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MTU-EC-OT-1-182/60
Record Dates: First submitted 2019-11-30; First posted 2019-12-06 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: ACL; screw fixation; graft inclination; reconstruction
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anterior cruciate ligament normal (Placebo Comparator): normal Anterior cruciate ligament reconstruction
  Interventions: Procedure: Interference screw
- Anterior cruciate ligament reconstruction (Experimental): Anterior cruciate ligament reconstruction and Position screw fixation
  Interventions: Procedure: Interference screw

INTERVENTIONS:
Procedure: Interference screw — Anterior cruciate ligament reconstruction (anterior screw fixation or posterior screw fixation)

SUMMARY:
The anatomic ACL reconstruction aims at functional restoration of the ACL to its native dimensions, collagen orientation and insertion sites. Even if the anatomic foot prints are correctly chosen for the tibial and femoral tunnels does the position of interference screw in the tibial tunnel alter the ACL orientation? The study hypothesized that the position of interference screw in the tibial tunnel would alter the graft orientation in anatomic ACL reconstruction. The purpose of this study was to compare graft orientation and inclination angle with posterolateral and anteromedial interference screw position in tibial tunnel in aperture fixation techniques.

ELIGIBILITY:
Inclusion Criteria:

* magnetic resonance imaging (MRI) of patients with ACL reconstruction was compared to MRI in which ACL was intact.
* patients with isolated ACL injury who underwent ACL reconstruction surgery using quadripled hamstrings graft and operated by a single senior surgeon
* Both pre-operative and post-operative MRI should be available for assessment
* No history of trauma in the post-operative or rehabilitation period

Exclusion Criteria:

* Concomitant bony or other ligament injury to the same knee
* history of previous surgery to the same knee
* Revision ACL reconstruction surgery
* surgery done at other center or by other doctors at our institute
* Pre-operative and/or post-operative MRI not available

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Inclination angle | 6 months
  Mean anterior cruciate ligament inclination angle in sagital x-ray (degree)

SECONDARY OUTCOMES:
post-operative complications | 6 months
  number of participants with revision, infection, reflex sympathetic dystrophy and re-rupture

IPD SHARING:
Plan to Share IPD: No